CLINICAL TRIAL: NCT00560963
Title: Combination of Antiangiogenic Therapy Using the mTOR-inhibitor RAD001 and Low Dose Chemotherapy for Locally Advanced and/or Metastatic Pancreatic Cancer - a Dose Finding Study
Brief Title: Treatment of Patients Suffering From a Progressive Pancreas Carcinoma With Everolimus (RAD001) and Gemcitabine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2491
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2012-11

CONDITIONS: Advanced or Metastatic Pancreatic Adenocarcinoma
Keywords: Advanced or metastatic pancreas carcinoma; gemcitabine; everolimus
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Everolimus

ARMS (1):
- 1 RAD001 (Experimental)
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus

SUMMARY:
A dose finding study in locally advanced and/or metastatic pancreatic cancer patients

ELIGIBILITY:
Inclusion criteria:

1. Histologically confirmed locally advanced, irresectable pancreatic adenocarcinoma (head, corpus, tail) with or without distant metastases
2. Adequate bone marrow, liver and renal function on everolimus treatment
3. At least one measurable lesion according to RECIST criteria that has not been previously irradiated.
4. Patients must be at least 4 weeks since prior major surgery and recovered, at least 2 weeks and recovered since prior minor surgery, completion of radiation, or completion of all prior systemic anticancer.
5. Age >18 years

Exclusion criteria:

1. Women who are pregnant or breast feeding.
2. Documented intolerance or history of allergy to everolimus or Gemcitabine.
3. History of another malignancy within 5 years prior to study entry, except curatively treated non-melanotic skin cancer or in-situ cervical cancer
4. Known or symptomatic central nervous system (CNS) metastases or leptomeningeal involvement
5. Chronic treatment with systemic steroids or another immunosuppressive agent
6. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus
7. Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumarin). Quick-value < 50 % or prothrombine time more than 1,5 fold higher

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of everolimus in combination with Gemcitabine | 8 weeks

SECONDARY OUTCOMES:
Safety & tolerability, pharmacokinetic assessments of Everolimus and Gemcitabine combination therapy in these patient populations. Phase II objective response rates (ORR), duration of response, progression-free survival (PFS), overall survival (OS) | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Germany (5):
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Merseburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Oberstaufen
  - Novartis Investigative Site, Ulm

REFERENCES:
- See also: Results for CRAD001C2491 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5163